CLINICAL TRIAL: NCT06974500
Title: Implementation of an Efferent Loop Stimulation Protocol Prior to Ileostomy Closure at La Paz University Hospital
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Luis Asensio Gomez, Consultant General Surgery, Hospital Universitario La Paz
Other Study IDs: PI-6255
Record Dates: First submitted 2025-04-24; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Ileus; Colorectal Cancer Control and Prevention; Stoma - Ileostomy
Keywords: Ileostomy , Stoma, Colorectal, Posoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Arm: Retrospective data from patients who did not undergo pre-ileostomy closure stimulation prior to the introduction of the efferent loop stimulation protocol.
- Arm Cases: Prospective patients with daily stimulation of the efferent loop at least two weeks prior to surgery with saline and thickener.
  Interventions: Procedure: Daily efferent limb stimulation for at least two weeks prior to surgery using saline solution and a thickering agent

INTERVENTIONS:
Procedure: Daily efferent limb stimulation for at least two weeks prior to surgery using saline solution and a thickering agent — Participants in the intervention group will undergo daily stimulation of the efferent limb for a minimum of two weeks prior to ileostomy closure. The procedure involves the instillation of a solution composed of saline and a thickening agent through the efferent limb of the ileostomy via the inactive orifice. This is performed by the patient at home following specific training and instructions provided during a preoperative consultation.
  The stimulation begins the day after the pre-anaesthesia consultation and is carried out once per day. Patients are supported with a structured follow-up, including one physical consultation in the stoma clinic, telephone contact with the research team every 48 hours, and access to an email address for queries. The objective of the intervention is to recondition the excluded colon before the restoration of intestinal continuity in order to reduce postoperative complications.
  Groups: Arm Cases

SUMMARY:
Stoma creation is a common surgical procedure, employed in certain contexts within general surgery, particularly in colorectal and emergency surgery. Although stoma formation is a life-saving technique, the diversion of intestinal contents has pathophysiological, aesthetic, and psychological repercussions on patients' lives. Stomas may be either permanent or temporary. In temporary cases, a second intervention is required to perform ileostomy closure and restore normal intestinal transit.

Several studies indicate that stimulation of the efferent loop prior to ileostomy closure yields benefits in patients' postoperative outcomes. Currently, there is no established protocol for this intervention at Hospital Universitario La Paz. However, implementing such a protocol-given that it is a simple, inexpensive, and accessible intervention-could offer significant cost-effectiveness. It may reduce complications and hospital stay, improve patients' quality of life, and represent a valuable contribution to the General Surgery Departmen

DETAILED DESCRIPTION:
Implementation of a Protocol for Efferent Limb Stimulation Prior to Ileostomy Closure at Hospital Universitario La Paz

The formation of stomas is a common surgical procedure, used in specific scenarios within general surgery, particularly in colorectal and emergency settings. While the creation of a stoma is often life-saving, the diversion of intestinal contents carries significant pathophysiological, aesthetic, and psychological repercussions for patients. Stomas may be permanent or temporary. In cases of temporary stomas, a second surgical procedure is required to close the ileostomy and re-establish normal intestinal continuity.

Several studies, as reviewed in this work, suggest that stimulation of the efferent limb prior to ileostomy closure provides measurable benefits in terms of patients' postoperative recovery. At present, however, there is no established protocol for this intervention at Hospital Universitario La Paz. This is despite its simplicity, low cost, and minimal risk, and its potential to improve patient outcomes, reduce postoperative complications, and shorten hospital stays. Implementing such a protocol could not only enhance patient care but also represent a meaningful quality improvement for the Department of General and Digestive Surgery.

The rationale behind this study is to demonstrate the clinical advantages of efferent limb stimulation before ileostomy closure and to establish a formal protocol for its use. This protocol would apply to patients with an ileostomy, regardless of the underlying condition, who are scheduled for intestinal reconstruction at Hospital Universitario La Paz. Complications following ileostomy closure are known to be common, often leading to prolonged hospitalisation. These complications result in increased direct costs from longer admissions, as well as additional use of healthcare resources through potential reoperations or pharmacological treatments.

Given these challenges, our objective is to reduce the duration of hospital stay and the incidence of complications by introducing a preoperative intervention that is both accessible and clinically effective. Efferent limb stimulation, conducted prior to closure, may provide an opportunity to mitigate common postoperative problems and improve overall patient recovery.

Our hypothesis is that stimulation of the efferent limb in patients with an ileostomy-using saline solution and thickening agents-administered between two and four weeks before intestinal reconstruction surgery, promotes faster recovery of bowel function, reduces length of hospital stay, and decreases postoperative complications. The primary outcome of interest is the reduction in the number of inpatient days, specifically measured from surgery to discharge.

Secondary objectives include evaluating the impact of the intervention on the incidence of postoperative paralytic ileus, diarrhoea, surgical site infections, and inflammatory response as indicated by C-reactive protein (CRP) levels. Additionally, the study will assess the feasibility and adherence to the newly implemented protocol.

The study is designed as a prospective cohort study with historical controls. The study population will consist of patients over the age of 18 with an ileostomy, regardless of the underlying pathology, who are scheduled for surgical restoration of intestinal continuity. Two groups will be analysed. The case group will include prospective patients who receive daily efferent limb stimulation with saline solution and a thickening agent for at least two weeks prior to surgery. The control group will consist of retrospective data from patients who underwent ileostomy closure prior to the implementation of this protocol and did not receive any form of preoperative stimulation.

Once enrolled, patients in the intervention group will follow the usual standards of care with the addition of the efferent limb stimulation protocol. All procedures and follow-up visits will be designed to ensure patient safety and will not introduce additional clinical risk

ELIGIBILITY:
IInclusion Criteria:

1. Subjects must be able to understand the purpose and risks of the study, provide informed consent, and authorise the use of confidential health information.
2. Patients over 18 years of age who, regardless of the underlying cause, have an ileostomy and a medical indication for intestinal transit reconstruction by a general surgeon.
3. Subjects who are able and willing to participate and to comply with follow-up for the duration of the study.

Exclusion Criteria:

1. Subjects with an ileostomy who do not wish to undergo intestinal reconstruction.
2. Subjects who are unable to complete at least two weeks of efferent loop stimulation prior to reconstruction surgery.
3. Subjects who do not provide consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who, regardless of the underlying cause, have an ileostomy and a medical indication for intestinal transit reconstruction.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
LOS | 30 days after reconstructive surgery
  Difference in mean number of days of hospital stay between control and case group

SECONDARY OUTCOMES:
Paralytic Ileus | Postoperative hospital stay (up to 15 days after surgery or until discharge, whichever occurs first)
  Percentage of patients diagnosed with paralytic ileus during admission in the case group compared to the control group
Diarrhoea | Postoperative hospital stay (up to 15 days after surgery or until discharge, whichever occurs first)
  Percentage of patients diagnosed with diarrhoea during admission in the case group compared to the control group
ISS | Postoperative hospital stay (up to 15 days after surgery or until discharge, whichever occurs first)
  Percentage of patients diagnosed with surgical wound infection 30 days after surgery in the case group compared to the control group
Protocol | through study completion, an average 2 years
  Percentage of the number of patients included in the protocol compared to the total number of ileostomies reconstructed since the protocol was implemented
CRP | Postoperative hospital stay (up to 15 days after surgery or until discharge, whichever occurs first)
  Percentage of the mean blood CRP value on the second and fourth day of patients undergoing EAE compared to the mean blood CRP value on the second and fourth day of patients without EAE.
PCT | Postoperative hospital stay (up to 15 days after surgery or until discharge, whichever occurs first)
  Percentage of the mean blood PCT value on the second and fourth posoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Luis Asensio, Consultant, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD due to privacy concerns and restrictions related to the informed consent provided by participants

REFERENCES:
- [Background] Fernandez Lopez F, Gonzalez Lopez J, Paz Novo M, Ladra Gonzalez MJ, Paredes Cotore J. Stimulation the efferent limb before loop ileostomy closure with short chain fatty acids. Cir Esp (Engl Ed). 2019 Jan;97(1):59-61. doi: 10.1016/j.ciresp.2018.06.018. Epub 2018 Oct 15. No abstract available. English, Spanish. PMID 30337046
- [Background] Lloyd AJ, Hardy NP, Jordan P, Ryan EJ, Whelan M, Clancy C, O'Riordan J, Kavanagh DO, Neary P, Sahebally SM. Efferent limb stimulation prior to loop ileostomy closure: a systematic review and meta-analysis. Tech Coloproctol. 2023 Dec 14;28(1):15. doi: 10.1007/s10151-023-02875-2. PMID 38095756
- [Background] Ocana J, Garcia-Perez JC, Labalde-Martinez M, Rodriguez-Velasco G, Moreno I, Vivas A, Clemente-Esteban I, Ballestero A, Abadia P, Ferrero E, Fernandez-Cebrian JM, Die J. Can physiological stimulation prior to ileostomy closure reduce postoperative ileus? A prospective multicenter pilot study. Tech Coloproctol. 2022 Aug;26(8):645-653. doi: 10.1007/s10151-022-02620-1. Epub 2022 May 21. PMID 35596903
- [Background] Garfinkle R, Demian M, Sabboobeh S, Moon J, Hulme-Moir M, Liberman AS, Feinberg S, Hayden DM, Chadi SA, Demyttenaere S, Samuel L, Hotakorzian N, Quintin L, Morin N, Faria J, Ghitulescu G, Vasilevsky CA, Boutros M; Bowel Stimulation Research Collaborative. Bowel stimulation before loop ileostomy closure to reduce postoperative ileus: a multicenter, single-blinded, randomized controlled trial. Surg Endosc. 2023 May;37(5):3934-3943. doi: 10.1007/s00464-022-09510-5. Epub 2022 Aug 19. PMID 35984521

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT06974500/Prot_SAP_000.pdf